CLINICAL TRIAL: NCT04706728
Title: "Receptive Music Intervention for the Abatement of Anxiety for In-patients Diagnosed With Unipolar Depression Who Receive Standard ECT Treatment". (ECT: Electroconvulsive Therapy).
Brief Title: Music Listening to Lower Anxiety During ECT Treatment.
Acronym: MIECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Lars Rye Bertelsen, External Lecturer, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VEK N-20200038
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Anxiety State
Keywords: Anxiety State; Unipolar Depression; Expert-Curated Playlists; ECT
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder | interventions — Rain; Lead

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT) with three arms, of which one is listening to playlists with sounds from nature for four weeks, one is listening to playlists with expert-curated music for four weeks, one is listening to playlists with expert-curated music for two weeks.
Masking Description: All participants are given a tablet with two playlists to choose from in each arm. Either two playlists with nature sounds, or two playlists with music.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Playlists with Expert-Curated Music - four weeks (Experimental): Patients can choose from two expert-curated playlists with music, matching the trajectory of the ECT treatment (immediately before-, during and after the procedure). Playlists are available to the patients for four weeks (the first eight ECT procedures).
  Interventions: Other: Listening to playlists with music prior to-, during and after the ECT procedure
- Playlists with Expert-Curated Music - two weeks (Active Comparator): Patients can choose from two expert-curated playlists with music, matching the trajectory of the ECT treatment (immediately before-, during and after the procedure). Playlists are available to the patients for two weeks (the first four ECT procedures).
  Interventions: Other: Listening to playlists with music prior to-, during and after the ECT procedure
- Playlists with Nature Sounds (Placebo Comparator): Patients can choose from two expert-curated playlists with recorded sounds from nature (Rain, Waves) during ECT treatment (immediately before-, during and after the procedure). Playlists are available to the patients for four weeks (the first eight ECT procedures).
  Interventions: Other: Listening to playlists with sound from nature (rain, waves) prior to-, during and after the ECT procedure

INTERVENTIONS:
Other: Listening to playlists with music prior to-, during and after the ECT procedure — Patients choose between two expert-curated playlists with music one day prior to ECT procedures for the first four weeks of their ECT treatment.
  Arms: Playlists with Expert-Curated Music - four weeks
Other: Listening to playlists with music prior to-, during and after the ECT procedure — Patients choose between two expert-curated playlists with music one day prior to ECT procedures for the first two weeks of their ECT treatment.
  Arms: Playlists with Expert-Curated Music - two weeks
Other: Listening to playlists with sound from nature (rain, waves) prior to-, during and after the ECT procedure — Patients choose between two expert-curated playlists with sounds from nature one day prior to ECT procedures for the first two weeks of their ECT treatment
  Arms: Playlists with Nature Sounds

SUMMARY:
The purpose of this study is to assess whether music listening is helpful in lowering anxiety in patients about to start their ECT treatment.

DETAILED DESCRIPTION:
In-patients at a psychiatric hospital referred to ECT treatment, is offered to participate in the study investigating whether listening to expert-curated playlists before-, during and after ECT treatment is helpful as a non-pharmacological intervention in lowering patients anxiety.

After written informed consent, participants will be randomised into two groups, one listening to playlists with music, one listening to sounds from nature (e.g. rain, ocean waves). Playlists will be administered by tablet+earphones in the waiting room, tablet+speaker in the room of procedure and tablet+bedside speaker in the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Capable in-patients of age at Aalborg University Hospital, Psychiatry - departments S7

  * S8, diagnosed with unipolar or bipolar depression, referred to ECT treatment.
* patients assessed to fit the study, by the head of departments S7 & S8
* Voluntary participation in the study after written informed consent.
* Patients can withdraw their consent at any point during the treatment trajectory.

Exclusion Criteria:

* Patients not compliant with the study, as assessed by head of departments
* Non-capable patients
* Patients who withdraw their written informed consent
* Patients using hearing aid
* Patients with former ECT treatment experience
* Patients who receive acute ECT Treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI-Y1) | First week of ECT treatment
  Measurement of patient anxiety before their first-, and before their second ECT procedure.
  Patients report of anxiety before their ECT treatment and therefore their anxiety is measured in validated STAI-Y1 questionnaire the evening before the first and before the second ECT procedure.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI-Y1) | First four weeks of treatment.
  Measurement of patient anxiety before their fifth.-, and before their ninth. ECT procedure.
  Patients report of anxiety before their ECT treatment and therefore their anxiety is measured in validated STAI-Y1 questionnaire during their first 8 ECT treatments, to see differences in anxiety levels over time (if any).

OTHER OUTCOMES:
Anxiety Symptom Scale questionnaire (ASS). | First four weeks of treatment.
  Defining the type of anxiety.
  Validated Anxiety Symptom Scale questionnaire (ASS), measured before 1st., 5th. and 9th. ECT procedure.
Non/validated questionnaire on patients experience of treatment quality. | First four weeks of treatment.
  Self-made questionnaire on patients' experience of the treatment quality using playlists as an add-on to Treatment As Usual (TAU).
Semi-structured Follow-Up interview. | One month after last ECT treatment
  Qualitative Follow-Up interview with two participants from each arm, approximately four weeks after their last ECT procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Lars R Bertelsen, Principal Investigator — Aalborg University, Doctoral Programme of Music Therapy.
Locations (1):
- Aalborg University Hospital, Psychiatry, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Collected data is solely used for publishing PhD. articles.